CLINICAL TRIAL: NCT01024205
Title: Upfront Sunitinib (SU011248) Therapy Followed by Surgery in Patients With Metastatic Renal Cancer: A Pilot Phase II Study [SuMR]
Brief Title: Sunitinib Malate Before and After Surgery in Treating Patients With Previously Untreated Metastatic Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barts and the London School of Medicine and Dentistry (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: OCTG-SuMR; CDR0000660317 (Registry Identifier: PDQ (Physician Data Query)); EUDRACT-2006-004511-21; REDA-4911; MREC-07/Q0603/58; PFIZER-OCTG-SuMR
Record Dates: First submitted 2009-12-01; First posted 2009-12-02 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2011-07

CONDITIONS: Kidney Cancer
Keywords: clear cell renal cell carcinoma; stage IV renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Sunitinib; Chemotherapy, Adjuvant; Neoadjuvant Therapy

INTERVENTIONS:
Drug: sunitinib malate
Other: laboratory biomarker analysis
Procedure: adjuvant therapy
Procedure: neoadjuvant therapy
Procedure: therapeutic conventional surgery

SUMMARY:
RATIONALE: Sunitinib malate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Giving sunitinib malate before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving sunitinib malate after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase II trial is studying how well giving sunitinib malate before and after surgery works in treating patients with metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine if neoadjuvant sunitinib malate can achieve a clinical benefit of 70% or more to the primary renal tumor prior to surgery and adjuvant sunitinib malate in patients with metastatic renal cancer.

Secondary

* Determine the time to radiological progression in these patients.
* Determine the overall survival of these patients.
* Determine the proportion of patients suitable for nephrectomy after neoadjuvant sunitinib malate.
* Determine the translational endpoints.

OUTLINE: Patients receive oral sunitinib malate once daily on days 1-28. Treatment repeats every 6 weeks for 3 courses. Approximately 2 weeks later, patients undergo a standard radical nephrectomy with lymph node dissection. Beginning at least 2 weeks after surgery, patients receive oral sunitinib malate on days 1-28. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.

Blood and tissue samples may be collected periodically for laboratory studies.

After completion of study treatment, patients are followed every 2 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed renal cell carcinoma

  * Measurable metastatic disease on CT/MRI imaging
  * Patients with suspicion of renal cancer on radiology must have a biopsy to confirm diagnosis of clear cell disease
* No prior therapy for renal cancer
* Judged by the treating physician to have the potential to derive clinical benefit from this treatment

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Absolute neutrophil count ≥ 1 x 10^9/L (without growth factor support)
* Platelet count ≥ 75 x 10^9/L
* Total bilirubin ≤ 2 times upper limit of normal (ULN) (except for patients with Gilbert disease)
* Serum creatinine ≤ 2 times ULN
* Serum transaminases < 5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 28 days after completion of study therapy
* Willing and able to comply with scheduled visits, treatment plan, and laboratory tests and other study procedures
* No congestive heart failure, myocardial infarction, or coronary artery bypass graft within the past 6 months, or ongoing severe or unstable arrhythmia requiring medication
* No other severe acute or chronic medical or psychiatric condition, or abnormal laboratory results that would impart, in the judgement of the investigator, excess risk associated with study participation or study drug administration or would make the patient inappropriate for entry into this study

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 7 days since prior and no concurrent potent CYP3A inhibitors, including any of the following:

  * Ketoconazole
  * Itraconazole
  * Clarithromycin
  * Erythromycin
  * Diltiazem
  * Verapamil
  * Delavirdine
  * Indinavir
  * Saquinavir
  * Ritonavir
  * Atazanavir
  * Nelfinavir
* At least 12 days since prior and no concurrent potent CYP3A inducers, including any of the following:

  * Rifampin
  * Rifabutin
  * Carbamazepine
  * Phenobarbital
  * Phenytoin
  * St. John's wort
  * Efavirenz
  * Tipranavir
* Concurrent radiotherapy allowed provided sunitinib malate is stopped one day before and resumed one day after radiotherapy
* Concurrent coumarin-derivative anticoagulants (e.g., warfarin) allowed (≤ 2 mg/day) for prophylaxis of thrombosis
* No concurrent treatment with a drug having proarrhythmic potential (i.e., terfenadine, quinidine, procainamide, disopyramide, sotalol, probucol, bepridil, haloperidol, risperidone, indapamide, or flecainide)
* No other concurrent investigational drug or participation in another clinical trial (unless approved by the sponsor)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2007-08; Primary Completion 2010-08 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Neoadjuvant sunitinib malate achieving a clinical benefit of ≥ 70%

SECONDARY OUTCOMES:
Time to radiological progression
Overall survival
Proportion of patients suitable for nephrectomy after neoadjuvant sunitinib malate

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Powles, MD, MRCP, Principal Investigator — Barts and the London School of Medicine and Dentistry
Locations (1):
- Orchid Clinical Trials Group at Barts and the London School of Medicine and Dentistry, London, England, United Kingdom

REFERENCES:
- [Result] Powles T, Chowdhury S, Bower M, Saunders N, Lim L, Shamash J, Sarwar N, Sadev A, Peters J, Green J, Boleti K, Augwal S. The effect of sunitinib on immune subsets in metastatic clear cell renal cancer. Urol Int. 2011;86(1):53-9. doi: 10.1159/000319498. Epub 2010 Oct 26. PMID 20975250
- [Derived] Stewart GD, Powles T, Van Neste C, Meynert A, O'Mahony F, Laird A, Deforce D, Van Nieuwerburgh F, Trooskens G, Van Criekinge W, De Meyer T, Harrison DJ. Dynamic epigenetic changes to VHL occur with sunitinib in metastatic clear cell renal cancer. Oncotarget. 2016 May 3;7(18):25241-50. doi: 10.18632/oncotarget.8308. PMID 27029034
- [Derived] Stewart GD, O'Mahony FC, Laird A, Rashid S, Martin SA, Eory L, Lubbock AL, Nanda J, O'Donnell M, Mackay A, Mullen P, McNeill SA, Riddick AC, Aitchison M, Berney D, Bex A, Overton IM, Harrison DJ, Powles T. Carbonic anhydrase 9 expression increases with vascular endothelial growth factor-targeted therapy and is predictive of outcome in metastatic clear cell renal cancer. Eur Urol. 2014 Nov;66(5):956-63. doi: 10.1016/j.eururo.2014.04.007. Epub 2014 May 10. PMID 24821582
- [Derived] Shaw GL, Hussain M, Nair R, Bycroft J, Beltran L, Green JS, Powles T, Peters JL. Performing cytoreductive nephrectomy following targeted sunitinib therapy for metastatic renal cell carcinoma: a surgical perspective. Urol Int. 2012;89(1):83-8. doi: 10.1159/000338057. Epub 2012 May 16. PMID 22614181